CLINICAL TRIAL: NCT03565341
Title: Evaluation of the Efficacy and Safety of the PiQo4 Picosecond Laser (PSL) System for the Treatment of Patients With Melasma: A Prospective, Randomized, Split Face Study Comparing the Added Value of 585nm Over 1064nm PSL
Brief Title: Efficacy and Safety of PiQo4 Device for Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Focus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Focus-PiQo4 Melasma-17-04
Record Dates: First submitted 2018-06-10; First posted 2018-06-21 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-02

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Face sides will be randomized to receive either 1064nm alone or 1064nm & 585nm combination treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Melasma (Experimental): Treatment of Melasma Using PiQo4 Laser System
  Interventions: Device: PiQo4

INTERVENTIONS:
Device: PiQo4 — PiQo4 Laser System for treatment of Melasma

SUMMARY:
Single center, Prospective, Open Label with Split-face Study Design. Face sides will be randomized to receive either 1064nm alone or 1064nm & 585nm combination treatment.

Each subject will receive up to 3 treatments at monthly intervals (±4 days). Follow-up visits will take place at 1, 3, and 6 months following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Female
2. Age= 18-75.
3. Fitzpatrick skin phototype = II-V
4. Melasma severity: diagnosed with mild to severe melasma lesions (MSS≥2)
5. Melasma type: Dermal or mixed type melasma, confirmed by Wood's lamp test
6. Melasma duration: The subject's melasma has persisted for greater than 6 months
7. Melasma previous treatments: has failed to respond to conventional treatment with hydroquinone or other topical lightening agents
8. Able to read, understand and provide written Informed Consent.
9. Able and willing to comply with the treatment/follow-up schedule and post treatment care
10. Agreed to use the same facial skin care products during the clinical trial period (including the follow-up period)
11. Agreed to the prohibition of the use of local/systemic corticosteroids or retinoids and other local/systemic lightening medications, and willing to abide by such instructions
12. Agreed to the daily use of an over SPF 50 sunblock on their face during the clinical trial period (including the follow-up period), and willing to abide by such instructions
13. Agreed to have their face photographed and willingness to allow Focus Medical (the study Sponsor) and Lumenis and the investigators to use de-identified photographs of the treated area for presentation and publication purposes
14. (In case of fertile women) Tested negative in the pregnancy test and agreed to use birth control contraceptives during the clinical trial period - Oral contraceptives are forbidden as they may influence the results of the clinical study.
15. Agreed not to undergo any other procedure on their face during their participation in the clinical trial

Exclusion Criteria:

1. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 3 months after completion of breastfeeding
2. Known hypersensitivity or contraindications to anaesthetic agents including lidocaine and its derivatives
3. Participation in a study of another device or drug within three months prior to enrolment or during the study.
4. Presence of open wounds or lesions in the area
5. Extensive scarring or tattoos in areas to be treated.
6. Having other pigmentation disorder
7. Having an excessive underlying vascular condition (e.g. dense network of capillaries).
8. Suffering from current or history of significant skin conditions in the treated area that could interfere with the evaluation (i.e. infection, dermatitis, or rash on their face) or requires the use of interfering topical or systemic therapy.
9. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
10. Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen
11. Subjects who are opposed to possible damage to the hair follicles with possible loss of hair in the treatment area
12. Laser or medium/deep chemical peel, or surgery, or filler treatments using collagen, hyaluronic acid, or any other material at area of treatment, within 6 months of initial treatment or during the course of the study.
13. IPL or superﬁcial chemical peel within the previous 1 month
14. Topical therapy with retinoids, imiquimod, 5-ﬂuorouracil, ingenol mebutate, diclofenac, alpha-hydroxy acids, or salicylic acids within the previous 1 month.
15. Currently using topical retinoid, hydroquinone or corticosteroid or whitening cream such as alpha arbutin, azelaic acid, kojic acid ascorbic acid or any cosmetics within 2 weeks
16. Lightening oral medication (hydroquinone, tranexamic acid), isotretinoid (or retinoid), light-sensitive medication, or steroids in the last 6 months
17. History of keloid scarring, hypertrophic scarring, or of abnormal wound healing.
18. History of connective tissue diseases such as systemic lupus erythematosus or scleroderma
19. Active leukoplakia, eczema, or psoriasis in the treatment area
20. History of post inflammatory pigmentary disorders, particularly a tendency for hyper- or hypo-pigmentation.
21. History of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis.
22. Has used photosensitizing drugs (e.g., Declomycin, sulfa antibiotics, phenothiazines, etc.) within a timeframe where photosensitization from these drugs may still be present
23. History of skin cancer in the treatment area
24. Significant concurrent illness or any disease state that in the opinion of the Investigator would interfere with the treatment or healing process
25. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
26. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician's discretion).
27. History of hormonal therapy in the last 3 months (e.g., estrogen, progesterone, or oral contraceptive)
28. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Percent of subjects having an improvement of at least 1 point on the MSS or ≥ 50% MASI score improvement on at least one of the face sides at the 1-month follow-up visit. | 1 month follow up
  The study will be deemed successful if the point estimate of the percent of successful subjects will be at least 50%.

SECONDARY OUTCOMES:
Percent of subjects having an improvement of at least 1 point on the MSS or ≥ 50% MASI score improvement on at least one of the face sides at the 3-month follow-up visit | 3 months follow up
Percent of subjects having an improvement of at least 1 point on the MSS or ≥ 50% MASI score improvement on each face side | 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: David J Goldberg, MD, Principal Investigator — Hackensack University Medical Center - Skin Laser & Surgery Specialists Of NY & NJ
Locations (1):
- Hackensack University Medical Center - Skin Laser & Surgery Specialists Of NY & NJ, Hackensack, New Jersey, United States